CLINICAL TRIAL: NCT06393179
Title: Epidemiology and Treatment Strategy of Open Respiratory Phenotype in Critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPEN-RESPIRATORY
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Mechanical Ventilation Pressure High; Critical Illness
Keywords: mechanical ventilation; airway closure; alveolar collapse
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P-V curve group (Experimental): Enrolled patients will receive a PV curve with a low-flow insufflation of 5 L/min starting from 0 cmH2O to a maximal airway pressure corresponding to the plateau pressure.
  Interventions: Other: pressure-volume curve with a low-flow insufflation of 5 L/min

INTERVENTIONS:
Other: pressure-volume curve with a low-flow insufflation of 5 L/min — The patient undergoes a pressure-volume curve with a low-flow insufflation of 5 L/min while in a state of analgesia, sedation, and absence of spontaneous breathing.

SUMMARY:
Monitoring airway pressure is essential for patients with mechanical ventilation. However, static airway pressure does not reflect alveolar pressure at all. Airway pressure is supposed to completely interrupt the communication between proximal airway opening and the distal alveolar and/or small airway structures. In this condition, some alveoli may still be inflated but do not communicate with proximal airways and auto-PEEP will give a biased estimated of mean alveolar pressure. To be note, distinguishing the airway closure and alveolar collapse can be challenging at times. The quasi-static PV curve is a useful bedside tool to set mechanical ventilation, which may help us to identify the airway closure and alveolar collapse. Meanwhile, the quasi-static PV curve can only reflects a global behaviour of the lung, while EIT may be a useful tool to assess the regional information on airway closure and alveolar collapse.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing controlled mechanical ventilation
* The duration of endotracheal intubation < 48 hrs

Exclusion Criteria:

* Severe hemodynamic instability
* Severe chronic lung disease requiring long-term home oxygen therapy
* Patients without analgesic sedation
* Decline to participate in the study
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
the rate of airway closure and alveolar collapse | up to 24 hours
  airway closure and alveolar collapse are monitored by PV curve with a low-flow insufflation of 5 L/min
Phenotype of respiratory open pressure | up to 24 hours
  According to the characteristics of the low inflation point of PV curve, the respiratory open pressure phenotype was constructed

SECONDARY OUTCOMES:
respiratory system compliance | up to 24 hours
  Respiratory system compliance is calculated as the ratio of tidal volume to the difference between plateau pressure and positive end-expiratory pressure.

CONTACTS AND LOCATIONS:
Overall Officials: ling liu, Principal Investigator — Zhongda Hospital
Locations (1):
- Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China